CLINICAL TRIAL: NCT07227623
Title: Randomized Trial of a Digital Health Intervention to Improve Physical Function and Wellness of Lung Cancer Survivors
Brief Title: A Digital Health Intervention to Improve Physical Function and Wellness of Lung Cancer Survivors
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Associate Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-529; RSG-24-1310262-01-CPHP (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-11-10; First posted 2025-11-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Advanced Lung Cancer; Physical Function
Keywords: Lung Cancer; Behavioral Intervention; Digital Health App; Physical Function
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROMOTE Digital Health App Intervention (Experimental): Patients will receive a study-issued tablet computer with the PROMOTE app that includes the following modules: 1) introductory education regarding the diagnosis and treatment trajectory of lung cancer; 2) behavioral interventions for improving physical function by managing fluctuations in energy and fostering engagement in valued life activities; 3) evidence-based breathing techniques for coping with dyspnea and improving lung function; 4) cognitive-behavioral strategies for enhancing sleep quality and efficiency; 5) approaches for increasing physical activity through adaptation and graded exercises; 6) tips for healthy eating and managing digestive side effects of cancer treatment, and 7) skills for managing mood symptoms through effective problem-, emotion-, and acceptance-based coping strategies. Patients will complete the intervention modules at their desired pace over approximately 10 weeks, in addition to their standard oncology care.
  Interventions: Behavioral: PROMOTE Digital Health App Intervention
- Enhanced Usual Care (Active Comparator): Patients will receive standard oncology care plus health educational materials about treatments for lung cancer, side effect management, and survivorship from the American Cancer Society (either in electronic or hardcopy formats).
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: PROMOTE Digital Health App Intervention — Patients will receive the PROMOTE digital health app, which includes educational modules focused on helping lung cancer survivors improve their physical function, management of breathlessness, sleep, physical activity, nutrition, and overall wellbeing.
  Arms: PROMOTE Digital Health App Intervention
Behavioral: Enhanced Usual Care — Patients will receive standard oncology care plus health educational materials about treatments for lung cancer, side effect management, and survivorship from the American Cancer Society (either in electronic or hardcopy formats).
  Arms: Enhanced Usual Care

SUMMARY:
The rationale for the proposed project is to improve the experience and outcomes of individuals diagnosed with lung cancer treated for cure. Survival rates in patients with stages I-III lung cancer continue to increase given progress in early detection and more effective treatments. However, the survivorship needs of this population are considerable and too often overlooked, especially with respect to their health behaviors, such as physical activity and nutrition, as well as persistent symptoms and side effects, including breathing difficulties and sleep disturbance. To ensure that as many patients as possible can access the information, support, and skills they require to navigate the diagnosis and treatment of lung cancer, the investigators worked with a multidisciplinary team to create a digital health intervention, called "PROMOTE." The investigators designed the PROMOTE mobile app for lung cancer survivors undergoing treatment to help them improve physical function, manage breathlessness and insomnia, increase physical activity, maintain a healthy diet, and enhance their overall wellbeing. To achieve the long-term goal to have PROMOTE become widely available to all lung cancer survivors, the next step in this research program is to conduct a randomized trial to demonstrate the benefits of the digital health intervention. Specifically, the investigators hypothesize that, compared to patients receiving enhanced usual care, those assigned to PROMOTE will report improved physical function, less difficulty with breathlessness and sleep disturbance, increased physical activity, healthier eating behaviors, fewer symptoms of anxiety and depression, and better quality of life. The investigators also plan to examine whether PROMOTE leads to more effective coping and greater confidence in patients' ability to manage their health (i.e., self-efficacy). For this project, the investigators will enroll lung cancer survivors receiving care at an academic cancer center and two affiliated community sites that provide care for diverse patient populations to ensure the results apply to a wide range of individuals with lung cancer. Participants will be randomly assigned either to receive the PROMOTE app intervention for 12 weeks or to an enhanced usual care control group that includes health education materials. Participants will complete surveys at enrollment and again at 6, 12, and 24 weeks after enrollment. At the end of the study, those assigned to the control group will be permitted to receive the PROMOTE app as well.

DETAILED DESCRIPTION:
Background: The population of lung cancer survivors continues to expand given advances in early cancer detection and cancer therapeutics significantly improving survival rates for these patients. However, interventions focused on survivorship are limited for those with lung cancer due to their historically poor prognosis. To address this unmet need, the investigators developed a digital health intervention, called "PROMOTE," for patients undergoing curative therapy for lung cancer to help them improve physical function, manage breathlessness and insomnia, increase physical activity, maintain a healthy diet, and enhance their overall wellbeing.

Objectives: The goal of the proposed study is to examine the impact of the PROMOTE mobile app intervention versus enhanced usual care (consisting of health education materials) on patient-reported outcomes in adults with non-small cell lung cancer (NSCLC) receiving treatment with curative intent that includes chemotherapy.

Study Aims: The specific aims are: 1) to evaluate the efficacy of PROMOTE versus enhanced usual care for improving patient-reported physical function (primary), dyspnea, sleep disturbance, physical activity, and eating behaviors; 2) to assess the efficacy of PROMOTE versus enhanced usual care for improving patient-reported self-efficacy, mood symptoms, and quality of life; and 3) to explore mediators and moderators of the effect of PROMOTE on patient-reported outcomes.

Study Design: The investigators will conduct a randomized controlled trial of PROMOTE versus enhanced usual care in 250 adult patients with stages I-III NSCLC receiving treatment with curative intent that includes chemotherapy. The investigators will examine the effect of the intervention on patient-reported physical function and other meaningful survivorship outcomes. Patients will be recruited from the Massachusetts General Hospital Cancer Center and two affiliated community sites. Participants will be randomized in a 1:1 fashion, stratified by study site and lung cancer treatment to ensure balanced representation between the two study groups on these factors. Patients assigned to PROMOTE will receive a tablet computer with instructions on how to use the digital app. Participants will complete self-report outcome measures at enrollment and again at 6, 12, and 24 weeks post-enrollment to evaluate the short and long-term impact of PROMOTE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of stage I-III non-small cell lung cancer
* Within six weeks of initiating treatment with curative intent that includes chemotherapy ± immunotherapy in the neo-adjuvant or adjuvant setting with surgery or as part of definitive chemoradiation
* Eastern Cooperative Oncology Group Performance Status = 0-2 (i.e., fully active to at least ambulatory and up and about more than 50% of waking hours)
* Ability to use a digital health intervention that includes verbal and written information in English
* Ability to complete questionnaires in English or Spanish
* Primary cancer care at one of the participating institutions

Exclusion Criteria:

* Significant uncontrolled psychiatric disorder or other co-morbid disease (e.g., dementia, cognitive impairment), which the treating oncology clinician reports would prohibit the patient's ability to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Physical Function | 12 weeks
  To compare patient-reported physical function at 12 weeks using the PROMIS Physical Function 8b Short Form, which is an 8-item measure that evaluates self-perceived capability of one's upper extremities, lower extremities, and activities of daily living (total scale score range: 8-40), with higher scores indicating better functioning.

SECONDARY OUTCOMES:
Patient-reported Dyspnea | 12 weeks
  To compare patient-reported dyspnea using the PROMIS Dyspnea Severity 10a Short Form, which is a 10-item measure that assesses the severity of shortness of breath or difficulty breathing in response to various specific activities (total scale score range: 0-30), with higher scores indicating worse dyspnea.
Patient-reported Sleep Disturbance | 12 weeks
  To compare patient-reported sleep disturbance at 12 weeks using the PROMIS Sleep Disturbance 8a Short Form, which is an 8-item measure that evaluates difficulties with sleep onset, maintenance, and quality (total scale score: 8-40), with higher scores indicating greater sleep disturbance.
Patient-reported Exercise and Eating Behaviors | 12 weeks
  To compare patient-reported exercise and eating behaviors at 12 weeks using the Simple Lifestyle Indicator Questionnaire, which is a 12-item measure that assesses multiple health behavior and wellness domains including physical activity, diet, alcohol use, smoking, and stress level (total score range: 0-10), with higher scores indicating a healthier lifestyle.

OTHER OUTCOMES:
Patient-reported Self-Efficacy | 12 weeks
  To compare patient-reported self-efficacy at 12 weeks using the PROMIS Self-Efficacy for Managing Daily Activities 4a Short Form, which is a 4-item measure that evaluates a person's confidence in their ability to perform various activities of daily living (total scale score range: 4-20), with higher scores indicating greater self-efficacy.
Patient-reported Anxiety Symptoms | 12 weeks
  To compare patient-reported anxiety symptoms at 12 weeks using the Hospital Anxiety and Depression Scale-Anxiety Subscale, which is a 7-item measure of anxiety symptoms (total subscale score range: 0-21), with higher scores indicating worse anxiety.
Patient-reported Depression Symptoms | 12 weeks
  To compare patient-reported depression symptoms at 12 weeks using the Hospital Anxiety and Depression Scale-Depression Subscale, which is a 7-item measure of depression symptoms (total subscale score range: 0-21), with higher scores indicating worse depression.
Patient-reported Quality of Life | 12 weeks
  To compare patient-reported quality of life at 12 weeks using the Functional Assessment of Cancer Therapy-Lung questionnaire, which is a 36-item measure of physical, social, emotional, and functional wellbeing as well as lung-cancer specific symptoms (total scale score range: 0-144), with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States